CLINICAL TRIAL: NCT05930431
Title: Physical Activity Variety's Impact on Physical Activity Participation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: U_of_Minnesota_PA_Variety
Record Dates: First submitted 2023-05-12; First posted 2023-07-05 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Physical Inactivity
Keywords: variety; consistency; HIIT (High intensity interval training); intervention; physical activity participation; enjoyment; motivation
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Two distinct physical activity groups occurring at the same time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity variety intervention (Experimental): Participants in the variety condition will be sent the link to their condition's website via email. The variety website will contain nine distinct high intensity interval training (HIIT) videos. The videos will be 30-minutes containing a five-minute warm-up, 20-minute workout, and a five-minute cool down. The website will emphasize the importance of having variety in one's physical activity routine. This will include reminders to have variety in selected workouts and the benefits associated with doing so. This emphasis will be supported through the counseling sessions provided to participants in the variety condition.
  Interventions: Behavioral: Physical activity variety intervention
- Physical activity consistency comparison condition (Active Comparator): Upon the completion of randomization, participants in the consistency condition will be sent the link to their condition's website via email. The consistency website will contain one HIIT video. The video will be 30-minutes and include a five-minute warm-up, 20-minute workout, and a five-minute cool down. The website will emphasize the importance of having consistency in one's physical activity routine. This will include reminders to be consistent in workouts and the benefits associated with doing so (Guiney & Machado, 2013). This emphasis will be supported through the counseling sessions provided to participants in the consistency condition.
  Interventions: Behavioral: Physical activity consistency comparison condition

INTERVENTIONS:
Behavioral: Physical activity variety intervention — The counseling in the variety condition will serve many purposes. The first session will concentrate on informing participants on the importance of having variety in their physical activity routine and how to access the variety of physical activities available to them. The variety condition will be instructed to complete at least three different HIIT workouts per week. They will be encouraged to complete more than three workouts. The following counseling sessions will be provided to not only continue supporting variety in physical activity but also to support participants' basic psychological needs.
  Arms: Physical activity variety intervention
Behavioral: Physical activity consistency comparison condition — The counseling in the consistency condition will serve many purposes. The first session will concentrate on informing participants the importance of having consistency in their physical activity routine and how to access the HIIT workout available to them. The consistency condition will be instructed to complete the provided HIIT workout three times per week. They will be encouraged to complete more than three workouts. The following counseling sessions will be provided to not only continue supporting consistency in physical activity but also to support participants' basic psychological needs.
  Arms: Physical activity consistency comparison condition

SUMMARY:
The primary purpose of the proposed study is to examine the effect of a home-based physical activity variety intervention on objectively measured physical activity in an eight-week randomized intervention trial.

DETAILED DESCRIPTION:
The primary purpose of the proposed study is to examine the effect of a home-based physical activity variety intervention on objectively measured physical activity in an eight-week randomized intervention trial. Early research on physical activity variety has observed increased physical activity participation, motivation, and enjoyment as a result of physical activity variety. However, previous studies examining variety have not included home-based interventions, objective measures of physical activity, or cardiovascular fitness classes.

Forty low-active college students will be randomly assigned to either an eight-week physical activity variety intervention (n=20) or a physical activity consistency comparison condition (n=20). Physical activity will be assessed via an accelerometer (e.g., Actigraph) at baseline and eight weeks, and psychosocial variables at baseline, four weeks, and eight weeks (i.e., post-intervention). Affect will be assessed at one, four, and eight weeks. Participants will receive counseling sessions and access to a website containing workouts appropriate to their condition.

ELIGIBILITY:
Inclusion Criteria:

* Engaged in no or low levels of physical activity (less than 90 minutes of moderate to vigorous intensity physical activity per week)
* Capable of completing a 30-minute session of physical activity
* 18-25 years of age old

Exclusion Criteria:

* Pregnant individuals
* Cannot read in English
* No access to the internet
* Healthcare providers have instructed them not to be active
* Any medical condition that would make physical activity unsafe or unwise

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Actigraph | Measuring the change from baseline to week 8.
  An electronic device worn on the right hip to identify motion.
Actigraph | Measuring the change from baseline to week 8.
  An electronic device worn on the right hip to identify steps taken.
Actigraph | Measuring the change from baseline to week 8.
  An electronic device worn on the right hip to identify energy expenditure.
Actigraph | Measuring the change from baseline to week 8.
  An electronic device worn on the right hip to identify time spent in different intensities of activity.
7-Day Physical Activity Recall Interview | Measuring change weekly from baseline until the eighth week of the intervention.
  Allows for tracking all bouts of MVPA that are at least 10 minutes in duration over the previous week. Physical activity is reported as minutes spent in moderate, hard, and very hard activities.

SECONDARY OUTCOMES:
Behavioral Regulation in Exercise Questionnaire (BREQ-2) | At baseline, weeks 4, and 8.
  Questionnaire: The BREQ-2 will assess participants' motivation regarding physical activity including amotivation, external regulation, introjected regulation, identified regulation, intrinsic regulation, and intrinsic motivation towards physical activity. The BREQ-2 is 19 items that includes a five-point Likert scale ranging from 0-4 with zero indicating "is not true" and four "very true." The BREQ-2 is a validated and commonly used measure examining SDT constructs.
Motives for Physical Activity Measure-Revised (MPAM-R) | At baseline, weeks 4, and 8.
  Questionnaire: The MPAM-R will be administered to assess participants' motives for physical activity. The five areas of motivation that are assessed include the following: Interest/enjoyment, competence, appearance, fitness, and social. Participants indicate how true an item is regarding why they engage in physical activity. Examples of the 30 items include, "It is fun," "I want to maintain physical strength for a healthy life," and "I like to be with others interested in this activity." The MPAM-R includes a Likert scale ranging from 1-7, with one indicating "not at all true" and a seven "very true." This measure has been validated for measuring motives for physical activity.
Psychological Need Satisfaction in Exercise (PNSE) | At baseline, weeks 4, and 8.
  Questionnaire: The PNSE will assess participants' satisfaction of their psychological needs, competence, autonomy, and relatedness. This measure is 18-items with six items examining each psychological need. An example of one item included for perceived competence is, "I feel that I am able to complete exercises that are personally challenging." An example of one item for perceived autonomy is, "I feel free to exercise in my own way." Lastly, one example of an item included for perceived relatedness is, "I feel attached to my exercise companions because they accept me for who I am." The items are scored using a Likert scale ranging from 1-6 with a one indicating "false" and a six representing "true." Higher values signify greater satisfaction of psychological needs. The PNSE has high reliability and is a commonly used measure for basic psychological needs.
Physical Activity Enjoyment Scale (PACES) | At baseline, weeks 4, and 8.
  Questionnaire: The PACES will assess participants' physical activity enjoyment. The PACES is an 18-item measure instructing participants to, "Measure how they feel about physical activity at this moment in time...." Participants rate each item using a Likert scale ranging from 1-7 with one and seven reflecting opposite ends of the spectrum. For example, the two anchors for the first item are, "I enjoy it" and "I hate it." In this example, a one aligns with "I enjoy it" and a seven aligns with "I hate it." Eleven of the items are reverse scored. Higher scores indicate higher levels of physical activity enjoyment. This measure has been found to be reliable and valid.
Bored of Sports Scale (BOSS) | At baseline, weeks 4, and 8.
  Questionnaire: The BOSS is a newly developed scale to assess boredom in physical activity. The BOSS is 11 items and includes a five-point Likert scale ranging from 0-4, with one representing "strongly disagree" and four representing "strongly agree." An example of an item is, "Exercising is dull and monotonous." Participants respond to prompts regarding their boredom in a specific bout of physical activity. This measure has been found to be reliable.
Exercise-Induced Feeling Inventory (EFI) | At baseline, weeks 4, and 8.
  Questionnaire: The EFI will assess exercise feeling. The 12-item questionnaire instructs participants to, "Indicate how each word describes how they feel at this moment in time...." Participants rate how they feel on a Likert scale of 0-4 with a zero indicating an item is "not felt;" whereas, a four indicates an item is "felt very strongly." Examples of the items are "refreshed," "worn out," and "energetic." The EFI is scored by summing the four subscales, which include revitalization, physical exhaustion, positive engagement, and tranquility. The four subscales each consist of three items. The EFI has demonstrated good internal consistency and reliability.
Feeling Scale (FS) | At weeks 1, 4, and 8.
  Questionnaire: The FS will assess affective valence experienced during physical activity. The FS is a two-item questionnaire that measures how participants are feeling and how much they are enjoying or enjoyed exercise. Participants rate their current feeling before, during, and after physical activity as part of the FS-current using a scale of -5 to +5, with a higher score indicating higher levels of positive affect. They rate their enjoyment as part of the FS-enjoyment on a scale of 1-7, with higher scores reflecting higher enjoyment. The FS is reliable for assessing in-exercise affect.

OTHER OUTCOMES:
Perceived Exercise Variety (PVE) | At baseline, weeks 4, and 8.
  Questionnaire: The PVE questionnaire will assess perceived variety of physical activity. Participants are asked to, "Please answer the following questions by considering how you typically feel while you are exercising." The questionnaire includes five items such as, "I feel like my exercise program is varied" and includes a 1-6 Likert scale with one indicating an item to be false and six indicating an item to be true. The PVE has been found to be valid and reliable.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
The Principal Investigator will be the only person with the authority to release the collected data. Confidential information will not be released under any circumstance. The original data file will stay in its original slate.

REFERENCES:
- [Background] Glaros, N. M., & Janelle, C. M. (2001). Varying the mode of cardiovascular exercise to increase adherence. Journal of Sport Behavior, 24(1).
- [Background] Juvancic-Heltzel JA, Glickman EL, Barkley JE. The effect of variety on physical activity: a cross-sectional study. J Strength Cond Res. 2013 Jan;27(1):244-51. doi: 10.1519/JSC.0b013e3182518010. PMID 22395266
- [Background] Sylvester BD, Standage M, McEwan D, Wolf SA, Lubans DR, Eather N, Kaulius M, Ruissen GR, Crocker PR, Zumbo BD, Beauchamp MR. Variety support and exercise adherence behavior: experimental and mediating effects. J Behav Med. 2016 Apr;39(2):214-24. doi: 10.1007/s10865-015-9688-4. Epub 2015 Nov 6. PMID 26546241